CLINICAL TRIAL: NCT02135666
Title: Long-term Hepatitis A and B Antibody Persistence in Healthy Adult Subjects, Primed 16 to 20 Years Earlier With GSK Biologicals' Combined Hepatitis A and B Vaccine, Twinrix® (SB208127) in Study HAB-084 (208127/084)
Brief Title: Evaluation of the Long-term Hepatitis A and B Antibody Persistence in Healthy Adult Subjects, Primed 16 to 20 Years Earlier With GSK Biologicals' Combined Hepatitis A and B Vaccine, Twinrix® (SB208127) in Study HAB-084 (208127/084)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: This study has been cancelled before initiation due to company's prioritisation decisions linked to resources restrictions.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 117307; 2013-004586-13 (EudraCT Number)
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Hepatitis B; Hepatitis A
Keywords: Twinrix; Long-term follow-up; Persistence; Hepatitis A; Antibody; Immunity; Hepatitis B; Combination vaccine; Adult
MeSH Terms: conditions — Hepatitis B; Hepatitis A | interventions — Blood Specimen Collection

ARMS (2):
- 2-dose Primed Group (Experimental): Adolescent subjects in this group received 2 doses of Twinrix Adult (720/20) (licensed as Ambirix in the EU) according to a 0, 6 months schedule in the primary study HAB-084 (208127/084).
  Interventions: Procedure: Blood sampling
- 3-dose Primed Group (Experimental): Adolescent subjects in this group received 3 doses of Twinrix Junior (360/10) according to a 0, 1, 6 months schedule in the primary study HAB-084 (208127/084).
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — At Years 16 - 20 after first dose of the primary vaccination in HAB-084 (208127/084) study.

SUMMARY:
The purpose of this study is to assess the long-term persistence of immunity to hepatitis A and B in adults who were vaccinated 16-20 years earlier with the combined hepatitis A and hepatitis B vaccine, Twinrix.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female who received two/three doses of Twinrix according to his/her group allocation in study HAB-084 (208127/084), and received no further dose of any hepatitis A and/or B vaccine since then.
* Written informed consent obtained from the subject.

Exclusion Criteria:

* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within six months prior to study entry. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs within six months prior to the study entry.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Administration of any hepatitis A and/or B vaccine at any time since completion of the primary vaccination series in HAB-084 (208127/084) study, including a challenge dose of the study vaccine, as a part of the study procedures, during the long-term persistence phase.
* Documented history of hepatitis A or B disease since completion of the primary vaccination series in HAB-084 (208127/084) study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Administration of immunoglobulins within six months prior to study entry.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity with respect to components of the study vaccine in terms of antibody titres | At each long-term follow-up (LTFU) visit (16-20 years after the first dose of primary vaccination)

SECONDARY OUTCOMES:
Occurrence of Serious adverse events (SAEs) | During the entire study period (Year 16-20)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hradec Králové, Czechia